CLINICAL TRIAL: NCT01502930
Title: MARI - Treatment of Nightmares Via the Internet - a Randomized Controlled Trial
Brief Title: Treatment of Nightmares Via the Internet
Acronym: MARI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICBT_Nightmares
Record Dates: First submitted 2011-12-22; First posted 2012-01-02 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Nightmares
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IRT (Experimental): Imagery Rehearsal Therapy
  Interventions: Behavioral: IRT
- CONT (Active Comparator): Stress reduction and positive imagery
  Interventions: Behavioral: Stress Reduction
- REG (No Intervention): Registration only

INTERVENTIONS:
Behavioral: IRT — Internet-based IRT with therapist support during 6 weeks
  Arms: IRT
Behavioral: Stress Reduction — Internet-based stress reduction with therapist support during 6 weeks
  Arms: CONT

SUMMARY:
This study is a randomized controlled trial (RCT) to evaluate the effect of an internet-based, guided self-help treatment of reoccurring and distressing nightmares. Imagery Rehearsal Therapy (IRT) will be compared to an active control treatment (CONT) and a recording-only group (REG). It is hypothesized that both active treatments will be superior to REG, and that IRT will be superior to CONT.

DETAILED DESCRIPTION:
Nightmares are distressing or frightening dreams, affecting 2.4 to 5% of the population. Suffering consists of disturbed sleep, fear and distress during night and/or day, expectancy anxiety and impaired functioning during the day.

Various forms of Cognitive Behavior Therapy (CBT) has been previously shown to be effective against nightmares and among them Imagery Rehearsal Therapy (IRT) has been the most promising. IRT consists of approaching the unpleasant dreams and to imagine a positive ending to them. So far IRT has been compared to untreated controls or treatments that have included methods to some extent similar to those in IRT, and it is therefore difficult to determine the specific effect of IRT.

Since access to CBT therapists is low, different types of self-help treatments for nightmares have been tested, but often these therapies have been provided without the assistance of a therapist, a procedure known to usually lower the effect of self-help treatments. So far, no nightmare treatment has been conducted over the Internet.

IRT will in this study be given as Internet CBT (ICBT) and will be compared to an active and credible control treatment (CONT) consisting of relaxation and exercise to focus on positive images or dreams, but without approaching or reinterpreting the nightmares. Relaxation Training has previously shown preliminary positive effects on nightmares. Both active treatments will be compared to a waiting list which only records how they manage their nightmares (REG).

The main purpose of this study is to examine whether the positive effects of IRT that has been seen in previous studies persists even when IRT is compared with a credible, active control treatment that does not contain the presumed active parts of the IRT. In addition, an untreated control group is used to ensure that the effects are not only due to spontaneous improvement. The control group will afterwards be treated with IRT without therapist support, in order to make a preliminary evaluation of the importance of therapist support.

Some researchers argue that nightmares are not to be seen only as something that is often caused or is a side effect of other conditions, but as a separate problem that should receive special treatment. Our study will help to determine whether it is possible to treat nightmares also in people with other problems such as posttraumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* have at least one nightmare (including awakening) or unpleasant dream (do not wake up) per week for at least a month.
* experience significant discomfort or distress due to nightmares/unpleasant dream.
* the content of the nightmares are not only related to a previous trauma.
* at least 18 years
* speaks, writes and read Swedish
* can not foresee any practical barriers to participation.

Exclusion Criteria:

* only suffers from night terrors and no nightmares according to criteria (a) to (c)
* has a high alcohol or drug use assessed by the AUDIT / DUDIT and assessment interview.
* somatic or psychiatric problems that are directly contraindicated or seriously hamper the implementation of the treatment (eg, psychotic disorders).
* have severe depression, defined as MADRS-S over 30 or suicidal risk judged by more than 4 points on the MADRS-S question 9 or according to the structured telephone assessment.
* has a total score over 76 on the IES-R (one standard deviation above the mean for individuals with a diagnosis of PTSD).
* is diagnosed with PTSD and can not provide proof that they have a current health care contact regarding PTSD.
* suffer from intrusive images or flashbacks during their waking hours (regardless of a PTSD diagnosis).
* currently undergoing some form of treatment that focuses on reducing symptoms of nightmares.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in nightmare frequency and distress | 6 weeks (Post) and 16 months (FU)
  Change (from baseline) of nightmare frequency and distress according to daily registrations

SECONDARY OUTCOMES:
Change (from baseline) in Nightmare Distress self-report | 6 weeks (Post) and 16 months (FU)
  Self-report of nightmare frequency and distress during last 14 days
Change (from baseline) in IES_R | 6 weeks (Post) and 16 months (FU)
  Impact of Events Scale, self-report to measure PTSD-symptoms
Change (from baseline) in ISI | 6 weeks (Post) and 16 months (FU)
  Insomni Severity Index, self-report to measure Insomnia symptoms
Change (from baseline) in MADRS-S | 6 weeks (Post) and 16 months (FU)
  Montgomery and Asberg Depressions Rating Scale - Self Report, to measure level of depression
Change (from baseline) in HADS | 6 weeks (Post) and 16 months (FU)
  Hospital Ancxiety and Depression Scale, self rating to measure anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Ph.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienehten (Internet Psychiatry Unit), Psykiatri Sydväst, SLSO, Stockholm, Sweden

REFERENCES:
- See also: The public page of the Internet-CBT treatment platform — http://www.internetpsykiatri.se